CLINICAL TRIAL: NCT07261449
Title: Effectiveness of Low-intensity Laser on Pain in Patients With Supraspinatus Tendinopathy. A Triple-Blind Randomized Controlled Trial.
Brief Title: Effectiveness of Low-intensity Laser on Pain in Patients With Supraspinatus Tendinopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia de Salamanca (Other)
Responsible Party: Principal Investigator, Jorge Velazquez, Principal Investigator, Universidad Pontificia de Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 221123
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Tendinopathy
Keywords: pain; range of motion; quality of life
MeSH Terms: conditions — Tendinopathy; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Experimental): Laser treatment on tendinophaty shoulder.
  Interventions: Device: Laser Group
- Placebo Group (Placebo Comparator): Placebo treatment on tendinophaty shoulder.
  Interventions: Device: Placebo Group

INTERVENTIONS:
Device: Placebo Group — A placebo treatment is carried out on the shoulder, simulating the application of the laser.
  Arms: Placebo Group
Device: Laser Group — Therapeutic laser treatment is performed on the shoulder.
  Arms: Laser treatment

SUMMARY:
Tendinopathy is an inflammatory process that occurs in and around the tendon when both are affected by a certain injury. In the case of the supraspinatus muscle it is one of the most frequent causes of shoulder pain. To test the efficacy of laser treatment in reducing shoulder pain caused by supraspinatus muscle tendinopathy. A randomized controlled clinical trial (RCT) was carried out in which a physiotherapy intervention was performed using therapeutic laser for three months, to observe the influence on the pain generated by supraspinatus muscle tendinopathy in the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Score of 3 or higher on the VAS scale for the shoulder.
* Adequate cognitive ability for comprehension.
* Rotator cuff tendinopathy confirmed by ultrasound at the study center, either due to tendon inflammation, presence of hypoechoic areas, calcification, fibrillar disorganization, and/or neovascularization in the supraspinatus muscle.
* Pain in the proximal lateral part of the arm that worsens with abduction.

Exclusion Criteria:

* Contraindications specific to laser treatment (e.g., tumors, presence of pacemaker or defibrillator, pregnancy, etc.).
* History of glenohumeral fracture and rheumatoid arthritis.
* Rheumatic, neurological, or structural polymyalgia affecting the joint.
* Previous surgeries.
* Pregnant or breastfeeding women.
* Taking anticoagulants or antiplatelet agents.
* Diabetes mellitus.
* Cardiac dysfunction.
* Infiltrative and/or rehabilitative treatment in the two months prior to recruitment.
* Pre-existing conditions associated with pain in the upper extremities. Difficulties with follow-up.
* Depression.
* Treatment with another intervention; during the study, they will not be able to undergo it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Pain | 3 months
  measured using the VAS scale, where 0 is the least possible pain and 10 is the greatest possible pain

SECONDARY OUTCOMES:
Range of motion | 3 months
  Shoulder mobility in the joint ranges of flexion, extension, abduction, adduction, and external and internal rotation. Measurement in degrees using a goniometer.
Patient quality of life | 3 months
  DASH questionnaire The score ranges from 0, which is equivalent to having no disability, to a maximum of 100, which is equivalent to having a very severe functional limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Redondo-Alonso L, Chamorro-Moriana G, Jimenez-Rejano JJ, Lopez-Tarrida P, Ridao-Fernandez C. Relationship between chronic pathologies of the supraspinatus tendon and the long head of the biceps tendon: systematic review. BMC Musculoskelet Disord. 2014 Nov 18;15:377. doi: 10.1186/1471-2474-15-377. PMID 25408141
- [Result] Haik MN, Alburquerque-Sendin F, Moreira RF, Pires ED, Camargo PR. Effectiveness of physical therapy treatment of clearly defined subacromial pain: a systematic review of randomised controlled trials. Br J Sports Med. 2016 Sep;50(18):1124-34. doi: 10.1136/bjsports-2015-095771. Epub 2016 Jun 10. PMID 27288517
- [Result] Romero-Morales C, Bravo-Aguilar M, Abuin-Porras V, Almazan-Polo J, Calvo-Lobo C, Martinez-Jimenez EM, Lopez-Lopez D, Navarro-Flores E. Current advances and novel research on minimal invasive techniques for musculoskeletal disorders. Dis Mon. 2021 Oct;67(10):101210. doi: 10.1016/j.disamonth.2021.101210. Epub 2021 Jun 4. PMID 34099238
- [Result] Asensio-Olea L, Leiros-Rodriguez R, Marques-Sanchez MP, de Carvalho FO, Maciel LYS. Efficacy of percutaneous electrolysis for the treatment of tendinopathies: A systematic review and meta-analysis. Clin Rehabil. 2023 Jun;37(6):747-759. doi: 10.1177/02692155221144272. Epub 2022 Dec 30. PMID 36583575
- [Result] Sanchez-Sanchez JL, Calderon-Diez L, Herrero-Turrion J, Mendez-Sanchez R, Arias-Buria JL, Fernandez-de-Las-Penas C. Changes in Gene Expression Associated with Collagen Regeneration and Remodeling of Extracellular Matrix after Percutaneous Electrolysis on Collagenase-Induced Achilles Tendinopathy in an Experimental Animal Model: A Pilot Study. J Clin Med. 2020 Oct 15;9(10):3316. doi: 10.3390/jcm9103316. PMID 33076550